CLINICAL TRIAL: NCT00400231
Title: The Fenofibrate and Metformin for Atherogenic Dyslipidemia (FAMA) Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 800860
Record Dates: First submitted 2006-11-09; First posted 2006-11-16 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Metabolic Syndrome x
Keywords: metabolic syndrome; Triglycerides; Insulin Resistance; inflammation; Cardiovascular Disease; Elevated triglycerides; without diabetes
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Inflammation; Cardiovascular Diseases; Hypertriglyceridemia | interventions — Fenofibrate; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Active Comparator): Metformin
  Interventions: Drug: Study Drug: Metformin
- 2 (Active Comparator): Fenofibrate
  Interventions: Drug: Study Drug: fenofibrate
- 3 (Active Comparator): Fenofibrate and Metformin
  Interventions: Drug: Study drugs: Metformin and fenofibrate
- 4 (Placebo Comparator)
  Interventions: Drug: Metformin and Fenofibrate placebo

INTERVENTIONS:
Drug: Study drugs: Metformin and fenofibrate — 145mg fenofibrate once/day and 2000mg/day of metformin for arm 3.
  Arms: 3
Drug: Study Drug: Metformin — 2000mg/day
  Arms: 1
Drug: Study Drug: fenofibrate — 145mg/day of fenofibrate
  Arms: 2
Drug: Metformin and Fenofibrate placebo — placebo metformin and fenofibrate
  Arms: 4

SUMMARY:
Patients with metabolic syndrome, insulin resistance, and elevated triglycerides of 150 mg/dl or higher will be randomized to one of four groups: 1) placebo; 2) metformin; 3) fenofibrate; or 4) combined metformin and fenofibrate for a period of 12 weeks after titration to target dose. We are interested in the effects of these therapies on triglyceride levels, HDL-C, insulin resistance, and markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

Subjects between the ages of 18 and 75 with both of the following risk factors:

1. Fasting triglycerides >= 150 mg/dl (but less than 800 mg/dl)
2. Glucose of 140 to 199 mg/dl, 2 hours after a 75 gm oral glucose load, a fasting HOMA level in the upper quartile (> 2.68), or a plasma triglyceride to high density lipoprotein cholesterol concentration > 3.0

And at least one of the following three:

1. Central obesity (waist size > 40 inches in men or >35 inches in women)
2. A systolic blood Pressure of >130 mmHg and/or a diastolic blood pressure of >85 mmHg and/or taking an antihypertensive medication.
3. HDL < 40 mg/dl for men or < 50 mg/dl for women

Exclusion Criteria:

1. Blood pressure > 180/95 mmHg (subjects may be re-screened after adequate blood pressure control has been obtained)
2. Women who are pregnant or lactating, or who are of child-bearing potential and not using an acceptable method of birth control.
3. Chronic renal insufficiency (serum creatinine >1.5 mg/dl in men and > 1.4 mg/dl in women
4. Any active liver disease or abnormal LFTs (>2x upper limit normal)(12)
5. Active infection, malignancy or chronic inflammatory disorder
6. Concomitant use of niacin, a bile acid sequestrant, or ezetimibe. If it is deemed safe by the patient's primary physician and by the principal investigator, patients may be screened for enrollment upon stopping these medications for at least 2 weeks.
7. Subjects on statins will need to be on less than maximal dose (e.g. < 80 mg per day for simvastatin or atorvastatin). Subjects will also need to have been on a stable dose of statin therapy for at least 1 month prior to enrollment and continue their currently prescribed statin at the same dose throughout the study. If it is deemed safe by the patient's primary physician and by the principal investigator, patients on maximal statin therapy (usually 80 mg/day) may reduce their dose of statin therapy to a sub maximal dose (usually 40 mg/day) for 4 weeks prior to screening for enrollment.
8. History of lactic acidosis(12)
9. Expected need for use of intravenous radiographic contrast during the study
10. More than moderate alcohol use (> 14 drinks per week)
11. Moderate to severe left ventricular dysfunction (ejection fraction <45%)
12. Decompensated heart failure or decompensated lung disease that has resulted in hypoxia or reduced peripheral perfusion within the past year regardless of left ventricular ejection fraction (thus patients with underlying heart disease, coronary artery disease, mild left ventricular dysfunction (ejection fraction > 45%), or lung disease that has been stable for at least one year will be eligible to participate)
13. Creatinine kinase (CK) levels ≥ 2.5 ULN or history of statin-induced myopathy. Patients with a CK level more than 2.5 times the upper limit of normal may undergo repeat testing up to two more times before being excluded (since vigorous physical activity can often elevate CK levels, and this would not increase the risk of myopathy).
14. Participation in an investigational drug study within 6 weeks prior to the screening visit
15. Surgery within the previous 30 days
16. Concomitant use of ketoconazole, itraconazole, cyclosporin A, erythromycin, or Clarithromycin.
17. Hemoglobin < 10 mg/dl, active use of coumadin, history of bleeding disorder, or abnormal clotting time (protime >14.6 seconds and aPTT > 37.0)
18. Septic shock
19. Acute coronary syndrome or stroke within 3 months prior to study
20. Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2005-08; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
triglyceride levels | 5 months

SECONDARY OUTCOMES:
HDL-C, Resistin, insulin resistance | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Frederick F. Samaha, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States